CLINICAL TRIAL: NCT00261547
Title: Pilot Study of Rituximab Treatment to Inhibit HLA Antibodies in Renal Allograft Recipients
Brief Title: Rituximab Treatment to Block HLA Antibodies in Renal Transplant Recipients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nina Tolkoff-Rubin, MD, Physician, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005p001524
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Chronic Rejection; Kidney Insufficiency
Keywords: Kidney transplantation; HLA
MeSH Terms: conditions — Renal Insufficiency | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental): this study has only one arm as the treatment group
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — All subjects will be treated with Rituximab 1000 mg (1 g) intravenously on days 1 and 15.
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine if administration of rituximab blocks the development of donor specific antibodies (DSA) in transplant recipients who have developed renal dysfunction and DSA after renal transplant. It is hoped that by blocking DSA production renal function will stabilize or improve.

DETAILED DESCRIPTION:
A long established risk factor for late renal allograft loss is the development of DSA. Recent studies from our group and others have shown that these antibodies are probably responsible for chronic rejection by attacking the vascular endothelium and fixing complement (detected as C4d in renal biopsies). Studies in humans and monkeys have shown that circulating antibody and complement deposition precede the development of chronic graft injury. Interruption of antibody production is a potential beneficial strategy to prevent late graft loss from this mechanism.

Therapeutic regimens that have been used in an attempt to deplete HLA or ABO antibodies include plasmapheresis, IVIg, tacrolimus and mycophenolate mofetil (MMF), and anti-CD20 (rituximab). Of these regimens, the most specific is anti-CD20, rituximab (rituxan), a therapy now FDA approved for B cell proliferative diseases. Although initially introduced for the treatment of neoplasm, the humoral immunosuppressant effects of rituximab have been shown to have clinical significance. Rituximab interferes with both primary and secondary humoral responses by eliminating B-cells prior to antigen exposure, thus interfering with differentiation into antibody secreting cells and specific antibody production.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a primary cadaver or living donor renal allograft
* 18-64 years of age
* At least 6 months and no more than 10 years post renal transplant
* Serum clearly positive for defined DSA
* Renal biopsy positive for C4d staining within 28 days before study Day 1 treatment
* Blood positive for Cd 19/20 cells at greater than/equal to 50 % of lower limit of normal
* Baseline serum creatinine 1.7-3.0 mg/dl
* On stable doses of tacrolimus and MMF for at least 1 month prior to study entry
* Able and willing to sign IRB approved consent form and comply with the requirements of the screen, treatment and follow-up phase of the protocol
* Negative serum pregnancy test (women of child bearing potential)
* Men and women of reproductive potential agree to use an acceptable method of birth control during treatment, for twelve months after treatment completion, or until B cell counts return to normal, whichever is longer

Exclusion Criteria:

* Hemoglobin: < 8.5 gm/dL
* Platelets: < 100.00/mm
* White blood cell count: < 3000/mm3
* AST or ALT . 2.5 x Upper Limit of Normal unless related to primary disease
* Positive Hepatitis B or C serology
* History of positive HIV
* Treatment with any investigational agen within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to study entry
* Previous treatment with rituximab (rituxan)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of recurrent infections
* Known active bacterial, viral, fungal, mycobacterial or other infection or any major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Ongoing use of high dose steroids (>10mg/day) or unstable steroid dose in the past 4 weeks.
* Lack of peripheral venous access
* History of drug, alcohol or chemical abuse within 6 months prior to screen
* Pregnancy or lactation
* Concomitant malignancies or previous malignancies
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac or pulmonary disease
* Any other disease, metabolic dysfunction, physical examination finding or clinical lab finding giving reasonable suspicion of disease or condition that contraindicates use of an investigational drug or that may affect the interpretation of the results or render subject a high rist from treatment complications
* Inability to comply with study and follow-up procedures

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Negative DSA by Luminex beads or ELISA | at 12 months post study medication
Lack of C4d deposition in peritubular capillary | on 12 month renal biopsy

SECONDARY OUTCOMES:
Renal allograft function: Serum creatinine, Calculated creatinine clearance, Urine protein, Urine protein-creatinine ratio | 12 months after study entry compared to the baseline
Change in chronic rejection pathology indices | on 12-month renal biopsy compared to baseline biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Tolkoff-Rubin, M.D., Principal Investigator — Massachusetts General Hospital